CLINICAL TRIAL: NCT06204081
Title: Exploration of the Short-term Effects and User Satisfaction of the Ceriter Stride One (CSO) Regarding the Prevention and Treatment of Freezing or Gait in Persons With Parkinson's Disease (pwP).
Brief Title: Short-Term Effect Of Ceriter Stride One (CSO) on FOG and Falling in pwP
Acronym: CSO_FOG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: ONZ - 2023 - 0501
Record Dates: First submitted 2023-12-01; First posted 2024-01-12 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Gait, Festinating; Parkinson Disease; Device Adherence
MeSH Terms: conditions — Gait Disorders, Neurologic; Parkinson Disease

STUDY DESIGN:
Intervention Model Description: One experimental group of pwP (H&Y stage 4, FOG) wear the sole a. 3 min. without using cues when FOG appears and b. 3 min. with using auditive cues when FOG appears. By randomisation of the conditions, the effect of cues on gait is studied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- persons with Parkinson's Disease, Hoehn & Yahr stage 4, FOG (Experimental): This group tests first without the use of cues (CSO evaluates gait pattern, but does not adjust), and then with cues.
  Interventions: Device: CSO_without cueing; Device: CSO_cueing

INTERVENTIONS:
Device: CSO_without cueing — The sole is worn without using the cueing application
Device: CSO_cueing — The sole is worn with using the cueing application

SUMMARY:
The Ceriter Stride One (CSO) is a "smart sole" with pressure sensors. The sole allows data on the displacement of the body's centre of gravity (COG), as well as spatiotemporal parameters, to be obtained via pressure recordings. Logarithms, released on the data captured by the sole, make it possible to recognise propulsion (forward movement of the CG), accompanied by a reduction in step length (festination) or feet remaining standing (freezing of gait). When the system registers incipient propulsion, an audio signal ("stop") is generated via an audio device and app on the mobile phone. The CSO aims to make the pwP stop before balance disturbance can occur, preventing further propulsion and falls.

The aim of the study is to explore the short-term effects of the CSO in terms of reducing (preventing) freezing of gait and fall risk in a pilot group of pwP whose functionality is limited (Hoehn and Yahr 4). Short-term impact on gait (episodes of freezing of gait, mean step length, mean gait speed) will be evaluated and user satisfaction surveyed.

DETAILED DESCRIPTION:
There is scientific evidence for making pwP stop at the onset of propulsion (when step length decreases and step frequency increases) in order to get the COG back within the base of support. Similarly, (auditory) cues are recommended to facilitate starting.

These principles are implemented with the CSO : the device makes the pmP stop at onset of propulsion and generates an auditory, rhythmic cue to facilitate starting and walking with larger steps (prevention).

This is an innovative application, not a standard-of-care intervention.

Protocol :

20 persons with Parkinson's disease (H&Y 4) (attending physical therapy at Movita).

The test proceeds in 3 stages : preparation / gait test / subjective evaluation :

Preparation

* Info / IC
* General data : age, sex, number of years since diagnosis, use of aids, medication, fall incidents last week (fall diary based on fall diary), (last intake) medication and current efficacy (VAS).
* MDS-UPDRS-II (degree of dependence), nFOGQ, Montreal Cognitive Assessment (MOCA).

Clinical gait test :

The soles are placed in the patient's shoes. If the patient uses an assistive device in daily life, the test is performed with an assistive device.

Following procedure is done in a randomized order*:

- Walking without auditory cue: for 3 minutes, the patient is asked to walk back and forth at a comfortable pace on a 4-meter course through a doorway (start : 2 meters before the doorway, stop : 2 meters beyond the doorway) without any auditory support. If no freezing occurs during this period, pwP is asked to turn 360° in the doorway.

The first 1.5 minutes gait is performed without a double task, the next 1.5 minutes with a cognitive double task (100 - 3 = ... - 3 = ... -3 = ...).

- Walking with auditory cues: for 3 minutes the patient is asked to walk back and forth at a comfortable pace along a 4-meter course through a doorway (start : 2 meters in front of the doorway, stop : 2 meters beyond the doorway) with auditory cues given at the occurrence of a freeze. If no FOG occured, the pwP is asked to turn 360° in the doorway.

The first 1.5 minutes gait is performed without a dual task, the next 1.5 minutes with a cognitive dual task (100 - 3 = ... - 3 = ... -3 = ...).

After each condition (with - without auditory cueing) a short break (2 minutes) is taken, during which a Borg scale for fatigue is taken. After the second condition, satisfaction with the effect of the aid is questioned (see below).

The entire gait test is filmed (by a 2nd person). In this way data, including the number of freezing episodes, can be checked.

*Randomization of conditions: per 2 patients. The first patient draws a card indicating whether or not the patient starts with auditory cues while walking. The 2nd patient then starts with the other condition, and so on. Thus we obtain 10 patients starting with the auditory cueing condition and 10 without.

Parameters considered : duration/step, gait asymmetry (pressure of left foot vs. right foot), number of freezing periods, distance walked, number of steps, mean step length.

Satisfaction questions

* On a scale of 1 to 10, how would you rate the level of comfort of the Ceriter Stride One?
* On a scale of 1 to 10, how safe do you feel when using the Ceriter Stride One?
* To what extent do you feel more secure, on a scale of 1 to 10, while walking by using the Ceriter Stride One?
* Open question : do you have any comments, concerns or questions of your own?

ELIGIBILITY:
Inclusion Criteria:

Parkinson's disease (or other Parkinsonism)

* gait impairment with freezing of gait (FOG)
* 18-80 years old
* I.C. (informed consent)
* Montreal Cognitive Assessment (MoCA) >25

Exclusion Criteria:

* unable to walk 4m without assistance
* MoCA < 25
* no FOG

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2023-12-05 (Actual); Primary Completion 2024-05-14 (Actual); Study Completion 2024-05-14 (Actual)

PRIMARY OUTCOMES:
The number of captured episodes with freezing of gait (FOG) | 2 times 3 minutes
  n (number of captured FOG-episodes : the less, the better)
The number of captured steps | 2 times 3 minutes
  n (number - more steps relate to a better mobility)
The difference between the pressure of steps with left versus right foot; as a measure of gait asymmetry. | 2 times 3 minutes
  mean presure data of left foot versus mean pressure data of right foot
mean step length | 2 times 3 minutes
  mean step length (cm)

SECONDARY OUTCOMES:
users satisfaction | after testing (5 min)
  comfort and safety of the tool are questioned on a scale of 1 to 10.

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Cambier, PhD, Principal Investigator — UGent, FGE
Locations (1):
- Ghent University, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zoetewei D, Herman T, Brozgol M, Ginis P, Thumm PC, Ceulemans E, Decaluwe E, Palmerini L, Ferrari A, Nieuwboer A, Hausdorff JM. Protocol for the DeFOG trial: A randomized controlled trial on the effects of smartphone-based, on-demand cueing for freezing of gait in Parkinson's disease. Contemp Clin Trials Commun. 2021 Jun 29;24:100817. doi: 10.1016/j.conctc.2021.100817. eCollection 2021 Dec. PMID 34816053
- See also: protocol of the DeFOG trial — https://pubmed.ncbi.nlm.nih.gov/34816053/